CLINICAL TRIAL: NCT06320301
Title: Evaluation of the Efficacy and Safety of Adebrelimab and a TKI in Combination With GEMOX in First-line Treatment of Advanced Biliary Tract Cancers (BTC): a Single-arm, Phase II Clinical Study
Brief Title: Adebrelimab and a TKI in Combination With GEMOX in First-line Treatment of Advanced Biliary Tract Cancers (BTC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-027-01
Record Dates: First submitted 2024-02-21; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Biliary Tract Cancer; Gemox Chemotherapy
Keywords: Biliary tract cancer; GEMOX; PD-L1; Adebrelimab; TKI
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — gemcitabine-oxaliplatin regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab + GEMOX + TKI (Experimental): Adebrelimab, 20 mg/kg, 30-minute intravenous infusion, once every 3 weeks (Q3W)
  TKI:
  Lenvatinib: 12 mg (3 capsules 4 mg) or 8 mg (2 capsules 4 mg) QD Apatinib: 250 mg orally, QD, 5 days on 2 days off or QOD Sorafenib: 0.4g (2 × 0.2g) twice or once daily Anlotinib: 12 mg orally before breakfast, QD. The drug was taken continuously for 2 weeks and stopped for 1 week.
  GEMOX:
  Gemcitabine 800mg/m2 and oxaliplatin 85mg/m2, IV, D2, D15, D29, until 6 cycles of treatment
  Interventions: Drug: Adebrelimab + GEMOX + TKI

INTERVENTIONS:
Drug: Adebrelimab + GEMOX + TKI — Adebrelimab 20 mg/kg, once every 3 weeks (Q3W), maintained for 1 year. The interval between two doses should not be less than 12 days.
  Tyrosine kinase inhibitor (TKI) Lenvatinib: 12 mg (3 capsules 4 mg) or 8 mg (2 capsules 4 mg) once daily (QD) at fixed times daily, on an empty stomach or with food; Apatinib: 250mg orally, QD, 5 days of medication, 2 days off (5 on 2 off) or once every other day (QOD), half an hour after meals; Sorafenib: 0.4g (2 × 0.2g) twice or once daily on an empty stomach or with a low-fat or medium-fat diet Anlotinib: 12 mg orally before breakfast, QD. The drug was taken continuously for 2 weeks and stopped for 1 week.
  GEMOX: gemcitabine 800mg/m2 and oxaliplatin 85mg/m2, intravenous infusion, D2, D15, D29, until 6 cycles of treatment were completed, or the patients who did not reach 6 cycles had intolerable adverse reactions, then the combination chemotherapy was terminated.
  Other Names: Adebrelimab+ tyrosine kinase inhibitor (TKI) + gemcitabine - oxaliplatin (GEMOX)

SUMMARY:
Patients with advanced biliary tract malignant tumors who had not received systematic treatment before and could not be cured were selected as the subjects of the study. The primary endpoint of the study was investigator-assessed 6-month progression-free survival (6-month PFS%) based on the RECIST v1.1 criteria, and 43 subjects were planned to be enrolled. Patients eligible for enrollment will receive Adebrelimab and a tyrosine kinase inhibitor (TKI) in combination with gemcitabine and oxaliplatin (GEMOX).

DETAILED DESCRIPTION:
This is an open-label, single-arm clinical study to observe and evaluate the efficacy and safety of Adebrelimab (PD-L1) and tyrosine kinase inhibitor (TKI) combined with gemcitabine and oxaliplatin (GEMOX) in the first-line treatment of patients with advanced biliary tract malignancies.

Subjects will be screened to receive Adebrelimab and TKI in combination with Gemcitabine and Oxaliplatin (GEMOX) after they are fully informed and sign the informed consent. Study treatment will continue until the subject develops intolerable toxicity, withdraws informed consent, and progresses as determined by the investigator in accordance with RECIST v1.1 (when the subject develops disease progression as defined in RECIST v1.1, if the investigator assesses that the subject continues to have clinical benefit and can tolerate the study treatment, The subject may continue treatment with the study drug; treatment may be terminated if the subject is no longer considered to have a clinical benefit), or other termination criteria specified in the protocol, whichever occurs first.

After the subjects were enrolled in the study, the safety visit will be conducted in D1 of each treatment cycle, and the safety visit and survival follow-up will be continued after the treatment.

Tumor imaging evaluation Imaging examination was performed every 6 weeks after enrollment to evaluate the efficacy. Additional imaging studies and evaluations may be performed at any time during the study if clinically indicated. Imaging evaluation of the tumor will continue until disease progression is confirmed by the investigator according to the RECIST v1.1 criteria or treatment is discontinued, whichever occurs later. Subjects who ended treatment for reasons other than investigator-confirmed disease progression (per RECIST v1.1) will also continue to be followed up at regular intervals for tumor imaging evaluation after the end of treatment.

If the subject withdraws the knowledge, has started other anti-tumor treatment (except Chinese patent medicine) or dies before the disease progression or termination of treatment confirmed by the investigator according to RECIST1.1 criteria, there is no need to continue the imaging evaluation. If the subject fails to meet the above termination criteria for imaging evaluation, the tumor efficacy evaluation of other efficacy evaluation criteria (RECIST v1.1, imRECIST) still needs to be continued even if the disease progression of a certain efficacy evaluation criteria occurs.

ELIGIBILITY:
Inclusion Criteria:

* 1) The patient voluntarily participated in the study and signed the informed consent;
* 2) ≥ 18 years old (calculated on the day of signing the informed consent), male or female;
* 3) Patients with advanced biliary tract malignant tumors confirmed by histopathology or cytology;
* 4) Subjects must be able to provide fresh or archived tumor tissue (formalin-fixed, paraffin-embedded [FFPE] blocks or at least 5 unstained FFPE slides) and their pathology reports. If less than 5 unstained slides are available from the subject or tumor tissue is not available (e.g., because of exhaustion of previous diagnostic tests), enrollment may be allowed on a case-by-case basis after discussion;
* 5) The subject is not suitable for surgery, or has progressed after surgery and/or local treatment;
* 6) Patients with progression after local therapy, where local therapy (including but not limited to surgery, radiotherapy, arterial embolization, arterial infusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection) has been completed at least 4 weeks prior to the baseline imaging scan, Toxicity (except alopecia) caused by topical treatment must be restored to the National Cancer Institute-Common Terminology Criteria for Adverse Events, Version 5.0 (NCI-CTCAE v5.0) rating ≤ 1;
* 7) No previous systemic therapy for BTC
* 8) At least one measurable lesion (according to the requirements of RECIST v1.1, the long diameter of the measurable lesion on spiral CT scan is ≥ 10 mm or the short diameter of the enlarged lymph node is ≥ 15 mm; the lesion that has received local treatment in the past can be used as the target lesion after the progress is confirmed according to the criteria of RECIST v1.1)
* 9) The physical condition score of the Eastern Cooperative Oncology Group (ECOG) was 0 ~ 2 (see Attachment 1 for the ECOG score standard);
* 10) Expected survival ≥ 12 weeks;
* 11) The functions of main organs are basically normal, and there are serious abnormalities of blood, heart, lung, liver, kidney, bone marrow and other functions and immunodeficiency diseases, which meet the requirements of the protocol: A) Blood routine examination: (except for hemoglobin, no blood transfusion within 14 days before screening, no use of granulocyte colony-stimulating factor [G-CSF], and no use of corrective therapy within 7 days) I. Hemoglobin ≥ 90 G/L; II. Neutrophil count ≥ 1.5 × 109/L; III. Platelet count ≥ 50 × 109/L; B) Biochemical examination: (no albumin transfusion within 14 days) I. Serum albumin ≥ 29 G/L; II. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN); III. Total bilirubin (TBIL) ≤ 1.5 times ULN;

IV. Creatinine Cr ≤ 1.5 X ULN or Cr clearance > 50 mL/min (Cockcroft-Gault formula below):

Male: Cr clearance = ( (140-age) × body weight)/ (72 × blood Cr) Female: Cr clearance = ( (140-age) × body weight)/ (72 × blood Cr) × 0.85 Weight unit: kg; Blood Cr unit: mg/mL; V. Urine protein < 2 + (if urine protein ≥ 2 +, 24-hour (H) urine protein can be quantified, and 24-hour urine protein < 1.0 G can be included in the group); C) Coagulation function: activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5 × ULN (can be screened for the use of stable dose of anticoagulant therapy such as low molecular weight heparin or warfarin and INR is within the expected therapeutic range of anticoagulant); D) Thyroid-stimulating hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be examined, and if T3 and T4 levels are normal, they can be included; Color Doppler echocardiography: left ventricular ejection fraction (LVEF) was greater than or equal to 60%.

* 12) Fertile women: must agree to abstain from sex (abstain from heterosexual intercourse) or use a reliable, effective method of contraception for at least 120 days from the signing of the informed consent until the final administration of the study drug. Serum HCG test must be negative within 7 days before the start of study treatment; And must be non-lactating. A woman is considered fertile if she has menstruated, has not yet reached postmenopausal status (no continuous periods for ≥12 months, no cause other than menopause is found), and has not undergone sterilization (such as hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).
* 13) For male patients whose partner is a woman of reproductive age, they must agree to abstain from sex for at least 120 days from the signing of the informed consent until the final administration of the study drug, or to use a reliable and effective method of contraception. Male subjects also had to agree not to donate sperm during the same time period. Male subjects with a pregnant partner are required to use condoms and do not need to use other methods of contraception.

Exclusion Criteria:

* 1) Active malignancies other than BTC within 5 years or at the same time. Cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc., could be included in the group.
* 2) Patients who are preparing for or have previously received organ or allogeneic bone marrow transplantation;
* 3) Other investigational drug treatment received within 28 days prior to the start of study treatment;
* 4) Moderate and severe ascites with clinical symptoms, i.e. requiring therapeutic puncture, drainage or Child-Pugh score > 2 (except for those with only a small amount of ascites on imaging but without clinical symptoms); uncontrolled or moderate or more pleural effusion and pericardial effusion;
* 5) If there is a history of gastrointestinal bleeding or a definite tendency of gastrointestinal bleeding within 6 months before the start of study treatment, such as bleeding risk or severe esophageal and gastric varices, local active gastrointestinal ulcer lesions, and persistent positive fecal occult blood, they should not be included in the group (if the fecal occult blood is positive at baseline, it can be reexamined, and if it is still positive after reexamination, Gastroduodenal endoscopy (EGD) is required, and esophagogastric varices with EGD suggesting a risk of bleeding are not eligible);
* 6) Abdominal fistula, gastrointestinal perforation, or abdominal abscess within 6 months prior to the start of study treatment;
* 7) Known presence of inherited or acquired bleeding (e.g., coagulopathy) or thrombophilia, e.g., in patients with hemophilia; current or recent (within 10 days prior to the start of study treatment) use of full-dose oral or injectable anticoagulants or thrombolytics for therapeutic purposes (low-dose aspirin, low-molecular-weight heparin, prophylactic use permitted);
* 8) current or recent use (within 10 days prior to study treatment) of aspirin (> 325 mg/day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel, and cilostazol;
* 9) Thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc., occurred within 6 months before the start of study treatment;
* 10) Clinical symptoms or diseases of the heart that are not well controlled, such as:

  1. LVEF (left ventricular ejection fraction) < 50% according to New York Heart Association (NYHA) standard II or above cardiac dysfunction or cardiac color Doppler ultrasound examination;
  2. unstable angina pectoris;
  3. Myocardial infarction within 1 year prior to the start of study treatment;
  4. Supraventricular or ventricular arrhythmias of clinical significance require treatment or intervention;
  5. QTc > 450ms (male); QTc > 470ms (female) (QTc interval is calculated by Fridericia formula; if QTc is abnormal, it can be detected three times at an interval of 2 minutes, and the average value is taken);
* 11)Hypertension that is not well controlled by antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg) (based on the average of BP readings obtained from ≥ 2 measurements) allows the use of antihypertensive therapy to achieve the above parameters; previous hypertensive crisis or hypertensive encephalopathy;
* 12) Major vascular disease (e.g., aortic aneurysm requiring surgical repair or with recent peripheral arterial thrombosis) within 6 months prior to the start of study treatment; severe, unhealed or dehiscent wounds, and active ulcers or untreated fractures; Major surgery has been performed within 4 weeks prior to the start of study treatment (except for diagnosis) or is expected to be performed during the study period;
* 13) There is evidence of intra-abdominal pneumatosis that cannot be explained by puncture or recent surgery;
* 14) prior or present central nervous system metastasis; Metastatic disease involving major Airways or vessels (for example, total occlusion of the main portal vein or vena cava due to tumor invasion, where the main portal vein is the confluence of the splenic vein and the superior mesenteric vein and where the hepatic portal vein divides into left and right branches) or a large mediastinal tumor mass located in the center (< 30 mm from the carina) should be excluded from the group;
* 15) Patients with history of hepatic encephalopathy; Current interstitial pneumonia or interstitial lung disease, or a previous history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or other pulmonary fibrosis, organizing pneumonia that may interfere with the judgment and management of immune-related pulmonary toxicity (e. Bronchiolitis obliterans), pneumoconiosis, drug-associated pneumonia, idiopathic pneumonia, or evidence of active pneumonia on computed tomography (CT) images of the chest during the screening period, or subjects with severely impaired lung function, with a history of radiation pneumonitis in the permissive field; active tuberculosis;
* 16) Active autoimmune disease or history of autoimmune disease with potential for recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [only subjects that can be controlled by hormone replacement therapy may be included]); Subjects with skin diseases that do not require systemic treatment such as vitiligo, psoriasis, alopecia, controlled type I diabetes mellitus on insulin therapy, or asthma that has completely resolved in childhood and does not require any intervention in adulthood may be included; asthma patients who require medical intervention with bronchodilators may not be included;
* 17) use of immunosuppressant or systemic hormone therapy for immunosuppression (dose > 10 mg/day prednisone or other iso-effective hormone) within 14 days prior to initiation of study treatment;
* 18) Known history of severe allergy to any monoclonal antibody drug;
* 19) Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia; therapeutic antibiotics administered orally or intravenously within 2 weeks prior to the start of study treatment (patients receiving prophylactic antibiotics (e.g., to prevent urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible for the study);
* 20) patients with congenital or acquired immune deficiency (such as HIV infection);
* 21) co-infection with hepatitis B and hepatitis C;
* 22) Have received live attenuated vaccine within 28 days prior to the start of study treatment or are expected to require such vaccine during treatment with or within 60 days of the last dose of Aderbelizumab In the judgment of the investigator, the patient has other factors that may affect the results of the study or lead to the forced termination of the study, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
the effectiveness of first-line treatment with Adebrelimab and a tyrosine kinase inhibitor (TKI) in combination with gemcitabine and oxaliplatin (GEMOX) in patients with advanced BTC | From enrollment to 6 months
  To evaluate the effectiveness of first-line treatment with Adebrelimab and a tyrosine kinase inhibitor (TKI) in combination with gemcitabine and oxaliplatin (GEMOX) in patients with advanced biliary tract cancer by assessing 6-month progression-free survival (6-month PFS%)

SECONDARY OUTCOMES:
To assess the progression-free survival (PFS) | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the effectiveness of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing progression-free survival (PFS).
To evaluate the time to progression (TTP) | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the efficacy and safety of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) in first-line treatment of patients with advanced biliary malignancies by assessing time to progression (TTP)
To evaluate the disease control rate (DCR), | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the effectiveness of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing disease control rate (DCR),
To evaluate the objective response rate (ORR) | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the effectiveness of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing objective response rate (ORR)
To evaluate the duration of response (DoR) | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the effectiveness of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing duration of response (DoR)
To evaluate the overall survival (OS). | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the effectiveness of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing overall survival (OS).

OTHER OUTCOMES:
To explore the correlation between biomarkers and the efficacy of the combination regimen. | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  Relationship between PD-L1 expression level in tumor tissue, PD-L1strong positive expression rate and the efficacy of Adebrelimab and TKI combined with gemcitabine-oxaliplatin (GEMOX)
The PFS based on an immunomodified RECIST (imRECIST） | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the efficacy of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing PFS based on an immunomodified RECIST (imRECIST）
The TTP based on an immunomodified RECIST (imRECIST） | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the efficacy of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing TTP based on an immunomodified RECIST (imRECIST）
The ORR based on an immunomodified RECIST (imRECIST） | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the efficacy of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing ORR based on an immunomodified RECIST (imRECIST）
The DCR based on an immunomodified RECIST (imRECIST） | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the efficacy of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing DCR based on an immunomodified RECIST (imRECIST）
The DoR based on an immunomodified RECIST (imRECIST） | From the date of enrollment until the date of the first documented progression or death from any cause, assessed up to 16 months after the enrollment of the last patient.
  To evaluate the efficacy of Adebrelimab and TKI in combination with gemcitabine and oxaliplatin (GEMOX) as first-line treatment for patients with advanced biliary malignancies by assessing DoR based on an immunomodified RECIST (imRECIST）

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No